CLINICAL TRIAL: NCT02308098
Title: Study Comparing Bronchodilator Efficacy of Two Dry Powder Inhalers, Budesonide/Formoterol Easyhaler and Symbicort Turbuhaler; a Randomised, Double-blind, Double-dummy, Multicentre, Single Dose, Crossover Study in Asthmatic Subjects
Brief Title: To Confirm Equivalent Bronchodilator Efficacy of the Test Product Compared to the Reference Product
Acronym: BUFODIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 3103013
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2015-06-30 (Estimated); Status verified 2015-01

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Budesonide; Budesonide, Formoterol Fumarate Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Budesonide/formoterol Easyhaler 320/9 ug/inhalation 4 inh (Experimental): Budesonide/formoterol Easyhaler 320/9 ug/inhalation 4 inh Placebo Symbicort Turbuhaler 320/9 ug/inhalation 4 inh
  Interventions: Drug: Budesonide/Formoterol Easyhaler 320/9 ug/inhalation 4 inh; Drug: Placebo Symbicort Turbuhaler 320/9 ug/inhalation 4 inh
- Budesonide/formoterol Easyhaler 320/9 ug/inhalation 1 inh (Experimental): Budesonide/formoterol Easyhaler 320/9 ug/inhalation 1 inh Placebo Symbicort Turbuhaler 320/9 ug/inhalation 1 inh
  Interventions: Drug: Budesonide/Formoterol Easyhaler 320/9 ug/inhalation 1 inh; Drug: Placebo Symbicort Turbuhaler 320/9 ug/inhalation 1 inh
- Symbicort Turbuhaler 320/9 ug/inhalation 4 inh (Experimental): Symbicort Turbuhaler 320/9 ug/inhalation 4 inh Placebo Budesonide/formoterol Easyhaler 320/9 ug/inhalation 4 inh
  Interventions: Drug: Symbicort Turbuhaler 320/9 ug/inhalation 4 inh; Drug: Placebo Budesonide/Formoterol Easyhaler 320/9 ug/inhalation 4 inh
- Symbicort Turbuhaler 320/9 ug/inhalation 1 inh (Experimental): Symbicort Turbuhaler 320/9 ug/inhalation 1 inh Placebo Budesonide/formoterol Easyhaler 320/9 ug/inhalation 1 inh
  Interventions: Drug: Symbicort Turbuhaler 320/9 ug/inhalation 1inh; Drug: Placebo Budesonide/Formoterol Easyhaler 320/9 ug/inhalation 1 inh

INTERVENTIONS:
Drug: Budesonide/Formoterol Easyhaler 320/9 ug/inhalation 4 inh
  Arms: Budesonide/formoterol Easyhaler 320/9 ug/inhalation 4 inh
Drug: Budesonide/Formoterol Easyhaler 320/9 ug/inhalation 1 inh
  Arms: Budesonide/formoterol Easyhaler 320/9 ug/inhalation 1 inh
Drug: Symbicort Turbuhaler 320/9 ug/inhalation 4 inh
  Arms: Symbicort Turbuhaler 320/9 ug/inhalation 4 inh
Drug: Symbicort Turbuhaler 320/9 ug/inhalation 1inh
  Arms: Symbicort Turbuhaler 320/9 ug/inhalation 1 inh
Drug: Placebo Symbicort Turbuhaler 320/9 ug/inhalation 4 inh
  Arms: Budesonide/formoterol Easyhaler 320/9 ug/inhalation 4 inh
Drug: Placebo Budesonide/Formoterol Easyhaler 320/9 ug/inhalation 4 inh
  Arms: Symbicort Turbuhaler 320/9 ug/inhalation 4 inh
Drug: Placebo Budesonide/Formoterol Easyhaler 320/9 ug/inhalation 1 inh
  Arms: Symbicort Turbuhaler 320/9 ug/inhalation 1 inh
Drug: Placebo Symbicort Turbuhaler 320/9 ug/inhalation 1 inh
  Arms: Budesonide/formoterol Easyhaler 320/9 ug/inhalation 1 inh

SUMMARY:
The purpose of this study is to confirm equivalent bronchodilator efficacy of the test product compared to the reference product.

ELIGIBILITY:
Main inclusion criteria:

* Written informed consent
* Asthma diagnosis for at least 6 months
* Prebronchodilator FEV1 45-90% of the predicted value
* Demonstration of reversible airway obstruction
* Stable asthma on the same regular treatment for at least 4 weeks before the study
* Non-smoker for at least 6 months before the study

Main exclusion criteria

* Respiratory infection within 4 weeks before the study
* Smoking history of more than 10 pack-years
* Other severe chronic respiratory disease than asthma
* Concurrent illness that would interfere with the interpretation of the study results or constitute a health risk for the patient if he/she takes part in the study
* Corrected QT interval > 450 ms in males or > 470 ms in females
* Abnormal serum potassium value or other clinically significant laboratory finding
* Systolic blood pressure over 180 mmHg and/or diastolic blood pressure over 100 mmHg
* Treatment with a long-acting β2-agonist, a xanthine-derivative, a β-blocker or with a corticosteroid (other than inhaled) within 4 weeks before the study
* Use of drugs that prolong QT-interval
* Women who are pregnant, breast-feeding or without reliable contraception
* Participation in another clinical drug study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-12; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Average FEV1 | 12 h
  FEV1 determined from serial spirometry and calculated on the basis of area under the curve

SECONDARY OUTCOMES:
Maximum FEV1 | 12 h
  Maximum FEV1 over the 12-hour serial assessments
FEV1 at 12 h | 12 h
  FEV1 at 12 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Hristo Metev, MD, Principal Investigator — Specialized Hospital for Active Treatment for Pneumophthisiatric Diseases Dr Dimitar Gramatikov-Ruse EOOD
Locations (1):
- Specialized Hospital for Active Treatment for Pneumophthisiatric Diseases Dr Dimitar Gramatikov-Ruse EOOD, Rousse, Bulgaria

REFERENCES:
- [Derived] Lahelma S, Vahteristo M, Metev H, Taseva M, Stamatova N, Bartha A, Schlezak J, Sairanen U. Equivalent bronchodilation with budesonide/formoterol combination via Easyhaler and Turbuhaler in patients with asthma. Respir Med. 2016 Nov;120:31-35. doi: 10.1016/j.rmed.2016.09.016. Epub 2016 Sep 25. PMID 27817813